CLINICAL TRIAL: NCT00804765
Title: Impact of Pregnant Women Education in Case of Overweight or Obesity on Risk of Child Overweight and Pregnancy Outcome
Brief Title: Impact of Education During Pregnancy in Overweight Pregnant Women
Acronym: ETOIG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AOM07093
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Overweight; Obesity; Pregnancy; Childhood Obesity
Keywords: Prevention; child obesity; pregnancy; overweight women; obese women
MeSH Terms: conditions — Overweight; Obesity; Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Therapeutic education
  Interventions: Other: Therapeutic education
- 2 (Placebo Comparator)
  Interventions: Other: Follow-up

INTERVENTIONS:
Other: Therapeutic education — Intensive training individual and collective teaching
  Arms: 1
Other: Follow-up — classical follow-up with two individual consultations
  Arms: 2

SUMMARY:
Metabolic environment of the foetus during pregnancy in obese women is altered and the child exposed at an increased risk of obesity. Rapid infancy and childhood weight gain is associated with subsequent obesity.

The purpose of the study is to test the efficacy of an educational intervention during pregnancy in obese or overweight women, on the reduction of rapid infancy weight gain in the two first years of life.

DETAILED DESCRIPTION:
In a first time, we propose to pregnant overweight women to participate a study based on the follow up of their pregnancy and of their child during the two first years of life. Women in agreement with the study sign a consent form and fill in a questionnaire about their quality of live.

We secondly randomized the women in two groups:

Group A: in this group an intervention is delivered. It provide education, at regularly scheduled sessions (20 weeks, 28 weeks, 35 weeks, and 2 month after delivering) and two dietary consulting. The sessions that stress about healthy eating and modest exercise assemble several women (no more than 10). Women in agreement with this intervention sign a consent form.

Group B: in this group, pregnant women are managed with standard care (at least one dietary consulting is proposed around 26 weeks).

Risk factors for child obesity are researched by questionnaire (parents smoking habit, mother and father level of education, family history of obesity, risk factors for gestational diabetes…). Mother weight measured at every clinic visit, is recorded as complications during pregnancy (HTA, preeclampsia, diabetes, fetal malformation …) and during delivery. Mother glycosylated haemoglobin is measured at birth.

Variables of interest for the children included at birth: gestational age, sex, neonatal pathology, hospitalisations and hypoglycaemia episode. Measurement, and method of infant feeding are recorded at birth, and by phone call every 2 months during 6 months, at 9 month, 1 year, 18 months and 2 years. At 4 months the mother fill in a questionnaire about the amount of milk or other foods eaten by the child.

A visit is planed at 2 years for:

* clinical examination of the child,
* recording of his nutritional and exercise habits
* questionnaire about quality of life of the mother and her health
* measurement of her BMI, arterial pressure, glycaemia before and after 75 g oral glucose-tolerance test, glycosylated hemoglobin, and lipid test.

ELIGIBILITY:
Inclusion criteria :

* Pregnant women who agree the study
* BMI > 25 kg/m². BMI is based on retrospective self reported weight of the patient before pregnancy.
* No more that 21 weeks of gestation.
* Social security

Exclusion criteria :

* women younger than 18 yrs,
* multiple gestation,
* high risk pregnancy,
* psychiatric pathology,
* diabetes diagnosed before the inclusion
* fetal malformation
* history of obesity surgery
* Women with no understanding of French language
* Women planning to move to another area.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2008-09; Primary Completion 2013-04 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
30 per cent reduction of rapid infancy weight gain at two years defined as > +0,67 change in weight SD score. The 0,67 SD represents the difference between the displayed centile lines on standard infant growth charts. | 30 Months

SECONDARY OUTCOMES:
-reduction of rapid infancy weight gain between 0 and 6 months | 30 months
-reduction of the number of children with BMI over 19 at 2 years | 30 months
-reduction of incidence of gestational diabetes, preeclampsia, HTA during pregnancy, caesarean, fetal macrosomia | 30 months
-reduction of spontaneous feeding at 4 months | 30 months
-increase of breastfeeding (number of women and duration) | 30 months
-reduction 1 and 2 years after pregnancy of mother weight and BMI (except second pregnancy) | 30 months
-reduction of abnormality of lipid and glycaemia test in women, 2 years after the pregnancy | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Sophie PARAT, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Necker, Paris, France

REFERENCES:
- [Result] Parat S, Negre V, Baptiste A, Valensi P, Bertrand AM, Chollet C, Dabbas M, Altman JJ, Lapillonne A, Treluyer JM, Elie C, Tauber M, Lorenzini F, Cosson E. Prenatal education of overweight or obese pregnant women to prevent childhood overweight (the ETOIG study): an open-label, randomized controlled trial. Int J Obes (Lond). 2019 Feb;43(2):362-373. doi: 10.1038/s41366-018-0205-z. Epub 2018 Sep 21. PMID 30242235